CLINICAL TRIAL: NCT06997640
Title: Comparative Analysis of Dynamic Stretching and Neural Mobilization Techniques on Pelvic Inclination in Early Middle-Aged Patients With Radicular Low Back Pain
Brief Title: Comparative Analysis of DS and NMT on Pelvic Inclination in Early Middle-Aged Patients With Radicular Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/826
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Stretching Protocol (Experimental)
  Interventions: Diagnostic Test: Dynamic Stretching Protocol
- Neural Mobilization Technique Protocol (Active Comparator)
  Interventions: Combination Product: Neural Mobilization Technique Protoco

INTERVENTIONS:
Diagnostic Test: Dynamic Stretching Protocol — Participants assigned to Group A will undergo a structured dynamic stretching protocol, designed to enhance lumbar flexibility, core muscle activation, and postural alignment, specifically targeting the pelvic inclination associated with radicular low back pain (RLBP). The intervention will be administered three times per week under the direct supervision of a qualified physiotherapist. Each session will last for 30 minutes, beginning with a 5-minute warm-up involving light aerobic activity such as marching or gentle trunk rotations to prepare the body for movement. This will be followed by 20 minutes of dynamic stretching exercises, focusing on the major muscle groups that influence pelvic and lumbar mobility.
  Arms: Dynamic Stretching Protocol
Combination Product: Neural Mobilization Technique Protoco — Participants in Group B will receive a standardized neural mobilization intervention, targeting the sciatic nerve and lumbar plexus, known to contribute to pain and restricted mobility in radicular low back pain (RLBP). The treatment will be conducted three times per week, with each session lasting 30 minutes under the guidance of an experienced physiotherapist trained in neurodynamic techniques. The session will begin with a 5-minute preparatory phase to position the participant comfortably and explain the sequence of movements. This will be followed by 20 minutes of gentle neural mobilization techniques, including nerve sliders and tensioners, performed through movements such as the Straight Leg Raise (SLR) sliders and the Seated Slump mobilization technique.
  Arms: Neural Mobilization Technique Protocol

SUMMARY:
Radicular low back pain (RLBP) is a common and debilitating condition characterized by nerve root irritation or compression, often resulting in altered biomechanics, muscular imbalances, and postural deviations such as anterior pelvic tilt.

DETAILED DESCRIPTION:
Rehabilitation strategies commonly focus on improving flexibility, neuromuscular control, and nerve mobility. Among these, dynamic stretching and neural mobilization techniques have shown individual effectiveness, but limited evidence exists on their comparative or combined effects on pelvic alignment and functional outcomes, particularly in early middle-aged adults. Addressing this gap could support the development of more targeted, evidence-based rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female
* Early middle-aged adults (aged 35-55 years)
* Diagnosed with radicular low back pain (RLBP) lasting more than 4 weeks
* Positive Straight Leg Raise (SLR) or Slump test
* Able to participate in physical therapy sessions 3 times/week(26)

Exclusion Criteria:

* History of spinal surgery or fractures
* Severe neurological deficits (e.g., foot drop, bladder/bowel dysfunction)
* Diagnosed with inflammatory or systemic conditions (e.g., ankylosing spondylitis, rheumatoid arthritis)
* Concurrent participation in other physical therapy programs
* Pregnant women or individuals with severe cardiovascular conditions

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
  The Visual Analog Scale (VAS) is a subjective but highly sensitive tool used for assessing pain intensity in clinical and research settings. It consists of a 10- centimeter horizontal line with endpoints labeled "0 = No pain" and "10 = Worst imaginable pain." Participants will be instructed to mark a point on the line that best reflects the intensity of their current pain, both at rest and during movement. The distance (in centimeters) from the "no pain" anchor to the marked point is then measured and recorded as the pain score.
Modified Schober Test | 12 Months
  It is a reliable and simple clinical method used to assess lumbar spine flexibility, particularly in the sagittal plane. It measures the extent of lumbar flexion by quantifying the increase in distance between two anatomical landmarks during forward bending. To perform the test, the examiner marks a point at the level of the posterior superior iliac spines (PSIS), which corresponds approximately to the L5 vertebra. A second mark is made 10 cm above and a third mark 5 cm below the initial point. The participant is then asked to bend forward as far as possible while keeping the knees straight.

CONTACTS AND LOCATIONS:
Locations (1):
- Private clinic Hyderabad Sindh, Hyderābād, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No